CLINICAL TRIAL: NCT03034252
Title: Retrospective Evaluation of Liposarcoma
Acronym: RELiSa
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Harrasser, Principal Investigator, Technical University of Munich
Other Study IDs: 448/11
Record Dates: First submitted 2017-01-22; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Survival , Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Patients with Liposarcoma — Evaluation of Liposarcoma treated in a single center

SUMMARY:
Retrospective Evaluation of Survival after Liposarcoma

ELIGIBILITY:
Inclusion Criteria:

* Patients with Liposarcoma treated surgically at our clinic

Exclusion Criteria:

* N/A

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Liposarcoma treated at our clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Survival rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: norbert harrasser, Principal Investigator — Klinikum rechts der Isar
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided